CLINICAL TRIAL: NCT05648500
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Safety, and Tolerability of Cenerimod in Adult Subjects With Moderate-to-Severe Systemic Lupus Erythematosus (SLE) on Top of Background Therapy
Brief Title: A Research Study to Evaluate the Effects of a New Oral Medicine Called Cenerimod in Adults With Systemic Lupus Erythematosus
Acronym: OPUS-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-064A301; 2022-002814-17 (EudraCT Number); 2024-515870-28-00 (EU CTIS Number)
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-08

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Musculoskeletal and connective tissue disorders; Connective Tissue Diseases; Immune System Diseases; Autoimmune Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Connective Tissue Diseases; Immune System Diseases; Autoimmune Diseases | interventions — cenerimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cenerimod 4 mg (Experimental): Participants will receive cenerimod once daily in addition to background SLE therapy.
  Interventions: Drug: Cenerimod
- Matching placebo (Placebo Comparator): Participants will receive matching placebo once daily in addition to background SLE therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cenerimod — Cenerimod will be supplied as a film-coated tablets at the dose of 4 mg.
  Other Names: ACT-334441
  Arms: Cenerimod 4 mg
Drug: Placebo — Matching placebo will be supplied as identical film-coated tablets formulated with the same excipients but without the active ingredient, cenerimod.
  Arms: Matching placebo

SUMMARY:
The goal of this clinical trial is to see how well cenerimod reduces symptoms of Systemic Lupus Erythematosus in adult patients with moderate to severe symptoms. The main questions it aims to answer are:

* How well cenerimod works on top of the treatment already being administered.
* How safe cenerimod is for adult patients with Systemic Lupus Erythematosus.

Researchers will compare one dose of cenerimod and a placebo to see how well cenerimod works when it is added to the treatment already being administered.

In this research study approximately 210 participants will receive cenerimod and approximately 210 participants will receive placebo for 12 months.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria at screening:

* Signed Informed Consent Form (ICF) prior to any study-mandated procedure.
* Diagnosis of Systemic Lupus Erythematosus (SLE) made at least 6 months prior to Screening, according to 2019 European League Against Rheumatism / American College of Rheumatology Criteria.
* A modified Systemic Lupus Erythematosus Disease Activity Index-2000 (mSLEDAI-2K) score ≥ 6 and clinical mSLEDAI-2K score ≥ 4 with at least 2 points for musculoskeletal or mucocutaneous manifestations (i.e., myositis, arthritis, rash, alopecia, mucosal ulcers). The mSLEDAI-2K score does not include "leukopenia".
* British Isles Lupus Assessment Group-2004 (BILAG) Grade B in ≥ 2 organ systems or a BILAG Grade A in ≥ 1 organ system.
* Physician's Global Assessment (PGA) score ≥ 1.0 on a 0 to 3 visual analog scale.
* Currently treated with one or more of the following SLE background medications:

  * Anti-malarials (≤ 400 mg/day hydroxychloroquine, ≤ 500 mg/day chloroquine, ≤ 100 mg/day quinacrine).
  * Mycophenolate mofetil (≤ 2 g/day) / mycophenolic acid (≤1.44 g/day).
  * Azathioprine (≤ 2 mg/kg/day).
  * Methotrexate (≤ 25 mg/week).
  * Oral Corticosteroids (OCS):

    * if OCS is the only SLE background medication: ≥ 7.5 mg/day and ≤ 30 mg/day prednisone or equivalent.
    * if OCS is not the only SLE background medication: ≤ 30 mg/day prednisone or equivalent.
  * Belimumab (≤10 mg/kg every 4 weeks intravenously [i.v.], or 200 mg/week subcutaneously [s.c.]).

Treatment with antimalarials, mycophenolate mofetil, mycophenolic acid, azathioprine, methotrexate or belimumab must have been started at least 90 days prior to Screening. Treatment with OCS must have been started at least 30 days prior to Screening.

• For women of childbearing potential (WoCBP):

* Negative serum pregnancy test at Screening.
* Agreement to undertake monthly urine pregnancy tests from Randomization up to 6 months after study treatment discontinuation.
* Agreement to use a highly effective method of contraception from Screening (Visit 1) up to 6 months after study treatment discontinuation.

Inclusion criteria at randomization:

* A clinical mSLEDAI-2K score ≥ 4 with at least 2 points for musculoskeletal or mucocutaneous manifestations (i.e., myositis, arthritis, rash, alopecia, mucosal ulcers).
* BILAG Grade B in 2 or more organ systems or a BILAG Grade A in 1 or more organ system.
* PGA score ≥ 1.0 on a 0 to 3 visual analog scale.
* Presence of at least one of the following biomarkers of serological evidence of active SLE (in a Screening sample as measured by central laboratory):

  * Anti-dsDNA antibodies elevated above normal,
  * Antinuclear antibodies with a titer of at least 1:160,
  * Anti-Smith antibody elevated above normal.
* Currently treated with one or more of the following SLE background medications that must be stable for at least 30 days prior to Randomization (except OCS, which must be stable for at least 15 days prior to Randomization):

  * Antimalarials (≤ 400 mg/day hydroxychloroquine, ≤ 500 mg/day chloroquine, ≤ 100 mg/day quinacrine);
  * Mycophenolate mofetil (≤ 2 g/day) / mycophenolic acid (≤ 1.44g/day);
  * Azathioprine (≤ 2 mg/kg/day);
  * Methotrexate (≤ 25 mg/week);
  * OCS:

    * if OCS is the only SLE background medication: ≥ 7.5 mg/day and ≤ 30 mg/day prednisone or equivalent.
    * if OCS is not the only SLE background medication: ≤ 30 mg/day prednisone or equivalent.
  * Belimumab (≤ 10 mg/kg every 4 weeks i.v. or ≤ 200 mg/week s.c.).
* WoCBP must have a negative urine pregnancy test at Randomization.

Main Exclusion Criteria:

* Pregnant, planning to be become pregnant up to Final Study Visit, or lactating women.
* Severe active central nervous system lupus or active severe or unstable neuropsychiatric SLE including but not limited to: aseptic meningitis; cerebral vasculitis; myelopathy; demyelination syndromes (ascending, transverse, acute inflammatory demyelinating polyradiculopathy); acute confusional state; impaired level of consciousness; psychosis; acute stroke or stroke syndrome; cranial neuropathy; status epilepticus; cerebellar ataxia; or mononeuritis multiplex:

  * That would make the subject unable to fully understand the ICF; OR
  * Where, in the opinion of the investigator/delegate, protocol-specified standard of care is insufficient and the use of a more aggressive therapeutic approach, such as adding i.v. cyclophosphamide and/or high dose i.v. pulse corticosteroid (CS) therapy or other treatments not permitted in the protocol is indicated.
* A diagnosis of mixed connective tissue disease or any history of overlap syndromes of SLE with psoriasis, rheumatoid arthritis, erosive arthritis, scleroderma, autoimmune hepatitis or uncontrolled autoimmune thyroid disease.
* History or presence of Mobitz type II or third-degree atrioventricular block, sick sinus syndrome, symptomatic bradycardia or syncope associated with cardiac disorders.
* Subjects who experienced myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack, vascular thrombosis, decompensated heart failure requiring hospitalization, or heart failure defined by the New York Heart Association Class III/IV within 6 months prior to Screening.
* Resting heart rate < 50 bpm as measured by the 12-lead ECG at Screening or at Randomization.
* An elevated QT interval corrected according to Fridericia's formula (QTcF) interval of > 470 ms (females) / > 450 ms (males) at Screening or at Randomization.
* History or presence of severe respiratory disease or pulmonary fibrosis, based on medical history, lung function, and chest X-ray (or CT scan as per local guidelines), performed at Screening or within 6 months prior to Screening.
* History of clinically relevant bronchial asthma or chronic obstructive pulmonary disease that has required treatment with oral or parenteral CS for more than a total of 2 weeks within the last 6 months prior to Screening.
* History or presence of malignancy (except for surgically excised and non-recurrent cutaneous basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma), lymphoproliferative disease, or history of total lymphoid irradiation within 10 years prior to Screening.
* Presence of any of the following abnormalities detected during the ophthalmological evaluation and/or by optical coherence tomography (OCT) during screening:

  * Macular edema of any cause: diabetic, cystoid, tractional.
  * Foveal degeneration, macular hole, macular pseudohole, hereditary or degenerative maculopathies.
  * Active uveitis, papilledema.
  * Retinal neovascularization of any cause and in any location.
* History of chronic liver or biliary disease (other than Gilbert's Syndrome) or subjects with alanine aminotransferase or aspartate aminotransferase > 3 × Upper Limit of Normal (ULN) or total bilirubin > 1.5 × ULN (unless in the context of known Gilbert's Syndrome).
* Significant hematology abnormality at screening assessment:

  * lymphocyte count < 500 /μL (0.5 × 10^9/L);
  * hemoglobin < 7 g/dL;
  * white blood cell count < 2000/μL (2.0 × 10^9/L); or
  * platelets < 25000/μL (25 × 10^9/L).
* Estimated glomerular filtration rate < 15 mL/min/1.73 m^2.
* Treatment with the following medications within 15 days or 5 half-lives of the medication (whichever is longer) prior to Randomization:

  * β-blockers, diltiazem, verapamil, digoxin, digitoxin, or any other anti-arrhythmic or heart-rate -lowering systemic therapy.
  * QT-prolonging drugs with known risk of torsade de pointes irrespective of indication.
* Treatment with the following medications within 30 days or 5 half-lives of the medication (whichever is longer) prior to Randomization:

  * Cyclophosphamide, cyclosporine, voclosporin, tacrolimus, sirolimus, etc.
  * Pulse methylprednisolone.
  * Vaccination with live vaccines (including live vaccines for COVID-19).
* Intra-articular, intramuscular or i.v. CS within 6 weeks prior to Randomization.
* Treatment with the following medications within 90 days or 5 half-lives of the medication (whichever is longer) prior to Randomization:

  * Leflunomide.
  * i.v. immunoglobulins.
* Treatment with any investigational agent within 90 days or 5 half-lives of the drug (whichever is longer) prior to Randomization.
* Treatment with B cell-depleting biological agents (e.g., rituximab or ocrelizumab) or biological immunosuppressive agents (e.g., anti-tumor necrosis factor [TNF], anti-interleukin [IL]-1, anti-IL6 therapies), within 12 months prior to Randomization.
* Treatment with anifrolumab within 6 months prior to Randomization.
* Treatment with any of the following medications any time prior to Screening:

  * Alemtuzumab,
  * Sphingosine-1-phosphate receptor modulators (e.g., fingolimod),
  * Subjects previously randomized to cenerimod or placebo in any trial involving cenerimod.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Response on Systemic Lupus Erythematosus Responder Index 4 (SRI-4) at Month 12 compared to baseline | At Month 12 compared to Day 1 (pre-dose baseline)
  Response on SRI-4 is defined as:
  * Reduction from baseline of at least 4 points in the modified Systemic Lupus Erythematosus Disease Activity Index-2000 score (mSLEDAI-2K [SLEDAI-2K modified to exclude leukopenia, thus mSLEDAI-2K]), and
  * No new British Isles Lupus Assessment Group-2004 (BILAG) A organ domain score and not more than one new BILAG B organ domain score compared to baseline, and
  * No worsening from baseline in subjects' lupus disease activity, where worsening is defined as an increase ≥ 0.30 points on a 3-point Physician's Global Assessment visual analog scale (PGA VAS), and
  * No violation of specified medication rules detailed in the core protocol.

SECONDARY OUTCOMES:
Response on BILAG-based Composite Lupus Assessment (BICLA) at Month 12 compared to baseline | At Month 12 compared to Day 1 (pre-dose baseline)
  Response on BICLA is defined as:
  * Improvement from baseline in disease activity as measured by BILAG. Improvement is defined as a reduction of all baseline BILAG A to B/C/D and baseline BILAG B to C/D and no BILAG worsening in other organ systems, where worsening is defined as ≥ 1 new BILAG A or ≥ 2 new BILAG B, and
  * No worsening from baseline in mSLEDAI-2K, where worsening is defined as an increase from baseline of > 0 points in mSLEDAI-2K, and
  * No worsening from baseline in the patient's lupus disease activity, where worsening is defined as an increase of ≥ 0.30 points on a 3-point PGA VAS, and
  * No discontinuation of investigational product, and
  * No violation of specified medication rules detailed in the core protocol.
Time to first confirmation of a 4-month sustained modified Systemic Lupus Erythematosus Disease Activity Index-2000 (mSLEDAI-2K) response | Day 1 (pre-dose baseline) to Month 12
  A response is defined as a reduction of at least 4 points from baseline.
Time to first confirmation of a 4-month sustained response in mucocutaneous manifestations (i.e., rash, alopecia, mucosal ulcers) | Day 1 (pre-dose baseline) to Month 12
  Response is defined as:
  * No increase in the overall mSLEDAI-2K score excluding mucocutaneous manifestations, and
  * Remission (score of zero) from baseline in the mSLEDAI 2K score of mucocutaneous manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (204):
- United States (29):
  - Providence Medical Foundation, Fullerton, California
  - California Research Institute, Huntington Park, California
  - University of Colorado Denver, Aurora, Colorado
  - RASF-Clinical Research Inc., Boca Raton, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Omega Research MetroWest, LLC, DeBary, Florida
  - SouthCoast Research Center, Inc., Miami, Florida
  - IRIS Research and Development, LLC, Plantation, Florida
  - Renew Health Clinical Research LLC, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Advance Quality Medical Research, Orland Park, Illinois
  - Accurate Clinical Research Inc. - Lake Charles, Lake Charles, Louisiana
  - Louisiana State University School of Medicine section of Rheumatology, New Orleans, Louisiana
  - Axon Clinical Research -Baltimore, Baltimore, Maryland
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - June DO, PC, Lansing, Michigan
  - Bronx Care Health and Wellness Center, The Bronx, New York
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Superior Clinical Reseach LLC, Smithfield, North Carolina
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Temple University Health Systems/ Lewis Katz School of Medicine, Philadelphia, Pennsylvania
  - Shelby Research, LLC, Memphis, Tennessee
  - Allen Arthritis, Allen, Texas
  - Accurate Clinical Research Inc., Baytown, Texas
  - Rheumatology Care Center, PLLC, Bellaire, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Houston MD Medspa and Wellness Clinic, Houston, Texas
  - Accurate Clinical Research Inc., Houston, Texas
  - Sun Research Institute, San Antonio, Texas
- Argentina (10):
  - Fundación Respirar, Buenos Aires
  - Instituto Medico CER, Buenos Aires
  - Aprillus Asistencia e Investigacion, Buenos Aires
  - Hospital Ramos Mejia, Buenos Aires
  - Arsema Clinica Adventista Belgrano, Buenos Aires
  - IR Medical Center /Hospital de Día/ Instituto de Reumatología y Traumatología, Mendoza
  - Instituto CAICI SRL, Rosario
  - Centro de investigaciones medicas Tucuman, San Miguel de Tucumán
  - Centro Integral de Reumatología, San Miguel de Tucumán
  - ICT (Investigaciones Clínicas Tucumán), San Miguel de Tucumán
- Brazil (13):
  - Santa Casa de Belo Horizonte, Belo Horizonte
  - Hospital Brasília, Brasília
  - Centro Mineiro de Pesquisas, Juiz de Fora
  - Instituto Méderi de Pesquisa e Saúde, Passo Fundo
  - Centro Multidisciplinar de Pesquisa Clínica (Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - LMK Servicos Medico S/S, Porto Alegre
  - IMPAR SERVICOS HOSPITALARES S/A ; Hospital São Lucas, Rio de Janeiro
  - SER - Serviços Especializados em Reumatologia da Bahia, Salvador
  - Hospital de Clínicas de Porto Alegre, Santa Cecília
  - Centro Multidiciplinar de Estudos Clínicos- CEMEC, São Bernardo do Campo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - CPClin - Centro de Pesquisas Clínicas, São Paulo
  - Ebserh Hospital de Clínicas da Universidade Federal de Uberlândia-HC-UFU, Uberlândia
- Bulgaria (9):
  - University Multi-profile Hospital for Active Treatment - Plovdiv AD, Plovdiv
  - "University Multiprofile Hospital for Active Treatment - Pulmed" OOD, Plovdiv
  - Medical Center ArtMed OOD, Plovdiv
  - Outpatient Clinic for Specialized Outpatient Medical Care - Medical Center Kyuchuk Parizh Ltd., Plovdiv
  - DCC 1 Ruse, Rousse
  - DCC-1-Sevlievo EOOD, Sevlievo
  - DCC "Sveta Anna" EOOD, Sofia
  - Acibadem City Clinic Diagnostic-Consultative Center" EOOD, 127 Okolovrasten pat, Mladost, Sofia
  - DCC Equita EOOD, Varna
- Colombia (10):
  - Clínica de la costa Ltda., Barranquilla
  - Bluecare salud SAS, Bogotá
  - IDEARG (Instituto de Enfermedades Autoinmunes Renato Guzmán), Bogotá
  - SERVIMED S.A.S Bucaramanga, Bucaramanga
  - Fundación Valle de Lili, Cali
  - Centro de Estudios de Reumatología y Dermatología, Cali
  - Preventive Care SAS, Chía
  - Hospital Pablo Tobón Uribe, Medellín
  - Fundación Centro De Excelencia En Enfermedades Crónicas No Transmisibles-FUNCENTRA, Montería
  - Healthy Medical Center SAS, Zipaquirá
- France (3):
  - Hôpital Pitié-Salpêtrière, Paris
  - CHU Félix Guyon Site Nord, Saint-Denis
  - CHU de Purpan, Toulouse
- Greece (9):
  - Naval Hospital of Athens, Athens
  - General Hospital of Athens "Hippokration", Athens
  - General Hospital of Athens "Laiko", Athens
  - University General Hospital "Attikon", Athens
  - General University Hospital of Larissa, Larissa
  - General University Hospital of Patras, Pátrai
  - Euromedica - Kyanos Stavros, Thessaloniki
  - General Hospital of Thessaloniki "Hippokration", Thessaloniki
  - 424 General Military Hospital, Thessaloniki
- India (10):
  - Sangini Hospital, Ahmedabad
  - Rajiv Gandhi Government General Hospital, Chennai
  - Nizam's Institute of medical Sciences, Hyderabad
  - Maharaja Agrasen Superspeciality Hospital, Jaipur
  - Radiance Hospital, Nagpur
  - Shree Hospital and Critical Care Centre., Nagpur
  - Assured Care Plus Hospital, Nashik
  - Coherence Pain & Arthritis Clinics, Pune
  - Vijaya Ortho & Trauma Centre, Sadashivnagar
  - Unity Hospital and Trauma Centre, Surat
- Japan (36):
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki-shi
  - National Hospital Organization Chiba Medical Center Chibahigashi National Hospital, Chiba
  - University of Yamanashi Hospital, Chuo-shi
  - St.Luke's International Hospital, Chūōku
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Hiroshima Prefectural Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Hitachi, Ltd. Hitachinaka General Hospital, Hitachi-Naka
  - National Kohnodai Medical Center, Japan Institute for Health Security, Ichikawa-shi
  - Tokai University Hospital, Isehara-shi
  - Kakogawa Central City Hospital, Kakogawa-shi
  - Shin-Kokura Hospital, Kitakyushu-shi
  - Kobe University Hospital, Kobe
  - Kobe City Medical Center General Hospital, Kobe
  - Kuwana City Medical Center, Kuwana-shi
  - Toho University - Ohashi Medical Center, Meguro-ku
  - University of Miyazaki Hospital, Miyazaki
  - Nagasaki University Hospital, Nagasaki
  - Chubu Rosai Hospital, Nagoya
  - Chukyo Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - IUHW Narita Hospital, Narita-shi
  - Niigata University Medical and Dental Hospital, Niigata
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - Ome Medical Center, Ome-shi
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - Japanese Red Cross Saitama Hospital, Saitama-shi
  - Sainokuni Higashiomiya Medical Center, Saitama-shi
  - Toho University Sakura Medical Center, Sakura-shi
  - Hokkaido University Hospital, Sapporo
  - National Hospital Organization Hokkaido Medical Center, Sapporo
  - Tohoku Medical and Pharmaceutical University Hospital, Sendai
  - Showa Medical University East Hospital, Shinagawa-ku
  - Tokyo Women's Medical University Hospital, Shinjuku-ku
  - Tomakomai City Hospital, Tomakomai-shi
  - Yokohama City Minato Red Cross Hospital, Yokohama
- Mexico (12):
  - Panamerican Clinical Research Mexico S.A. de C.V., Cuernavaca
  - Consultorio Privado de Especialidad, Guadalajara
  - Centro de Estudios de Investigación Básica y Clínica, S.C., Guadalajara
  - Consultorio Médico de Reumatología - Hospital Aranda de la Parra, León
  - Biológicos Especializados S.A. de C.V., Mexico City
  - CITER, Centro de Investigación y Tratamiento de las Enfermedades Reumáticas S.A. de C.V., Mexico City
  - Unidad de Atención Médica e Investigación en Salud, Mérida
  - Centro de Investigación Clínica Chapultepec S. A. de C. V., Morelia
  - SMIQ, S. de R.L. de C.V., Querétaro
  - Centro de Atención e Investigación Cardiovascular del Potosí, S.C., San Luis Potosí City
  - Unidad de Investigaciones Reumatológicas A.C, San Luis Potosí City
  - Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V., Zapopan
- Philippines (7):
  - Chong-Hua Hospital, Cebu City
  - Davao Doctors Hospital, Davao City
  - Mary Mediatrix Medical Center, Lipa
  - Makati Medical Center, Makati
  - UP-PGH, Manila
  - Far Eastern University - Nicanor Reyes Medical Foundation, Quezon City
  - Jose R. Reyes Memorial Medical Center, Santa Cruz
- Poland (9):
  - INTER CLINIC Piotr Adrian Klimiuk, Bialystok
  - Centrum Medyczne Pratia Częstochowa, Częstochowa
  - Centrum Medyczne Angelius Provita, Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Małopolskie Badania Kliniczne, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Velocity Nova Sp. z o. o., Lublin
  - Zespół Poradni Specjalistycznych REUMED, Lublin
  - Malwa-Med Iwona Chlebicka, Wroclaw
- Romania (6):
  - Neomed Brasov, Brasov
  - SC Sana Monitoring SRL, Bucharest
  - Delta Health Care SRL, Bucharest
  - Spitalul Clinic Dr. Ion Cantacuzino, Bucharest
  - Spitalul Clinic Judetean de Urgentã Craiova, Craiova
  - SC Medaudio-Optica SRL, Râmnicu Vâlcea
- South Korea (7):
  - Pusan National University Hospital, Busan
  - Catholic University of Daegu (Daegu Catholic University Medical Center), Daegu
  - Seoul National University Hospital, Junggu
  - Hanyang University Hospital, Seongdong-gu, Seoul
  - Ewha University Mokdong Hospital, Yangcheon-gu, Seoul
  - KonKuk University Medical Center, Gwangjin-gu, Seoul
  - Seoul Saint Mary's Hospital of the Catholic University of Korea, Seocho-gu, Seoul
- Taiwan (10):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - TRI-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan
- Thailand (9):
  - Vajira Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital (PMK), Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Division of Rheumatology, Chiang Mai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Songklanagarind Hospital, Songkhla
  - Fort Sunpasithiprasong Hospital, Ubon Ratchathani
- Ukraine (15):
  - Communal Non-Commercial Enterprise "Cherkasy Regional Hospital of Cherkasy Regional Council", Cherkasy
  - Communal Non-Commercial Enterprise "Khmelnytsky Regional Hospital" of Khmelnytsky Regional Council, Khmelnytskyi
  - Clinic of Modern Rheumatology, Kyiv
  - Kyiv City Clinical Hospital #3, Kyiv
  - Kyiv Railway Clinical Hospital #2 of Branch "Health Center" of Joint-Stock Company "Ukrainian Railway", Kyiv
  - State Ins Nat Scie Cen M.D.Strazhesko Ins of Cardio Clin, Kyiv
  - Communal Non-Commercial Enterprise of Kyiv Regional Council Kyiv Clinical Regional Hospital, Consultation and Diagnostic Center, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Com Non-Com Entr of Lviv Reg Coun "Lviv Reg Clin Hos, Rheu Dprt, Danylo Halytsky Lviv Nat Med Uni, Lviv
  - Medical Center of Limited Liability Company "Kalyna. Center of Modern Medicine, Lviv
  - Medical Centre "Academical Medical Group" LLC, Lviv
  - Uzhhorod City Multidisciplinary Clinical Hospital, Uzhhorod
  - Private Small-Scale Enterprise Medical Centre "Pulse", Therapeutical Department, Vinnytsia
  - Municipal Nonprofit Institution "Vinnytsia City Clinical Hospital #1", Vinnytsia
  - Communal Enterprise "Hospital #1" of Zhytomyr City Council, Consultation and Treatment Department "Scientific Research Center", Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Askanase AD, D'Cruz D, Kalunian K, Merrill JT, Navarra SV, Cahuzac C, Cornelisse P, Murphy MJ, Strasser DS, Trokan L, Berkani O. Cenerimod, a sphingosine-1-phosphate receptor modulator, versus placebo in patients with moderate-to-severe systemic lupus erythematosus (CARE): an international, double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Rheumatol. 2025 Jan;7(1):e21-e32. doi: 10.1016/S2665-9913(24)00246-7. Epub 2024 Nov 22. PMID 39586304